CLINICAL TRIAL: NCT02016898
Title: The Effect of Sponge Versus No-Sponge Placement of Mitomycin-C on the Outcomes of Trabeculectomy With Ex-PRESS Glaucoma Filtration Device
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00048136
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Results first posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open angle glaucoma; trabeculectomy; mitomycin-C; express mini-shunt
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sponge placement of Mitomycin-C (Experimental): Randomization will be stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Interventions: Procedure: Placement of the sponge; Drug: Mitomycin-C
- Irrigation placement of Mitomycin-C (Experimental): Randomization will be stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Interventions: Drug: Mitomycin-C

INTERVENTIONS:
Procedure: Placement of the sponge
  Arms: Sponge placement of Mitomycin-C
Drug: Mitomycin-C

SUMMARY:
The primary focus of this study is to assess intraocular pressure and complication rates between patients who receive mitomycin-C using a sponge versus no-sponge.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 years and older at screening.
2. Diagnosis of chronic angle-closure glaucoma or open-angle glaucoma, phakic or pseudophakic, with visual field or optic disc changes characteristic of glaucoma.
3. Suitable candidate for trabeculectomy with Ex-PRESS glaucoma filtration device with MMC in the superonasal quadrant in the study eye which the physician deems as medically necessary.
4. Capable and willing to provide consent

Exclusion Criteria:

1. Unable or unwilling to provide consent
2. Any previous ocular surgeries in the study eye preventing placement of the trabeculectomy with Ex-PRESS glaucoma filtration device with mitomycin-C in the superonasal quadrant
3. Any previous glaucoma drainage devices in the study eye
4. Any abnormality other than glaucoma in the study eye that could affect applanation tonometry.
5. Presence or history of any abnormality or disorder that could interfere with the study procedure or prevent the successful completion of the study.
6. Presence or history of uveitis within 10 years or any other ocular infection or inflammation within 14 days before day 1.
7. Any significant unstable cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
8. Known Pregnancy or Breastfeeding

   Physical and Laboratory Findings
9. Conjunctival scarring precluding a superonasal implantation location.
10. Vitreous in the anterior chamber.
11. Abnormality preventing reliable applanation tonometry in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Herndon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Quist MS, Brown N, Bicket AK, Herndon LW. The Short-term Effect of Subtenon Sponge Application Versus Subtenon Irrigation of Mitomycin-C on the Outcomes of Trabeculectomy With Ex-PRESS Glaucoma Filtration Device: A Randomized Trial. J Glaucoma. 2018 Feb;27(2):148-156. doi: 10.1097/IJG.0000000000000830. PMID 29189540

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were retroactively removed due to not satisfying the inclusion/exclusion criteria. An additional three subjects had uncertain group allocation due to clerical errors.
Groups:
- Sponge Placement of Mitomycin-C: Randomization stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Placement of the sponge
  Mitomycin-C
- Irrigation Placement of Mitomycin-C: Randomization stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Irrigation placement
  Mitomycin-C
Period: Overall Study
Arm/Group | Sponge Placement of Mitomycin-C | Irrigation Placement of Mitomycin-C
Started | 50 | 45
Completed | 45 | 40
Not Completed | 5 | 5
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sponge Placement of Mitomycin-C: Randomization will be stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Placement of the sponge
  Mitomycin-C
- Irrigation Placement of Mitomycin-C: Randomization will be stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Irrigation placement
  Mitomycin-C
- Total: Total of all reporting groups
Arm/Group | Sponge Placement of Mitomycin-C | Irrigation Placement of Mitomycin-C | Total
Number analyzed (Participants) | 50 | 45 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9.6) | 73.1 (8.3) | 70.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 26 | 16 | 42
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 45 | 95

OUTCOME MEASURES:

1. Primary Outcome: Complication Rates
Description: To assess complication rates between patients who receive mitomycin-C using a sponge versus irrigation
Time Frame: post-operative day 1 to month 6
Measure: Count of Participants; unit: Participants
Groups:
- Irrigation Placement of MMC: Randomization will be stratified by age (age ≥65 or age < 65), baseline IOP (IOP ≥ 28 mmHg or IOP < 28 mmHg), and concurrent cataract surgery.
  Irrigation placement
  Mitomycin-C
Arm/Group | Sponge Placement of Mitomycin-C | Irrigation Placement of MMC
Number analyzed (Participants) | 50 | 45
Participants | 29 | 28
Statistical Analysis 1: Comparison: Sponge Placement of Mitomycin-C vs Irrigation Placement of MMC; Test type: Other; p = 0.7, Chi-squared; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.67 to 1.29]

2. Secondary Outcome: Change in Intraocular Pressure
Description: To assess final intraocular pressure lowering between patients who receive mitomycin-C using a sponge versus irrigation
Time Frame: post-operative day 1 to month 6
Population: Five participants in each group were not included due to being lost to follow-up or deceased.
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Sponge Placement of Mitomycin-C | Irrigation Placement of MMC
Number analyzed (Participants) | 45 | 40
mmHg (millimeters of mercury) | -8.4 (1.6) | -8.2 (1.2)
Statistical Analysis 1: Comparison: Sponge Placement of Mitomycin-C vs Irrigation Placement of MMC; Test type: Other; p = 0.539, t-test, 1 sided; Median Difference (Final Values) = 0.2, Standard Deviation 2.01

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sponge Placement of Mitomycin-C | Irrigation Placement of Mitomycin-C
All-Cause Mortality (participants affected / at risk) | 1/50 | 1/45
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/45
Other Adverse Events (participants affected / at risk) | 29/50 | 28/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sponge Placement of Mitomycin-C (N=50) | Irrigation Placement of Mitomycin-C (N=45)
Cystic blebs (Eye disorders) | 8 | 5
Shallowing of anterior chamber (Eye disorders) | 1 | 3
Hypotony (Eye disorders) | 5 | 14
Choroidal effusion (Eye disorders) | 3 | 3
Suprachoroidal hemorrhage (Eye disorders) | 0 | 1
Hyphema (Eye disorders) | 1 | 1
Wound leak (Eye disorders) | 18 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes